CLINICAL TRIAL: NCT07041047
Title: Open Clinical Investigation to Evaluate Efficacy And Safety of the Medical Device "Apaisant Serum - Ingrown Nails" in The Treatment of Ingrown Nail
Brief Title: Evaluation of Apaisant Serum - Ingrown Nails for Ingrown Toenails
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Footcare Laboratories - Poderm Professional (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23E2009
Record Dates: First submitted 2025-03-17; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Ingrown Toenails; Ingrown Nail Inflammation
Keywords: Ingrown nails; Ingrown toenails treatment; Pain relief; Topical treatment; Medical device; Nail inflammation; Clinical study on ingrown nails
MeSH Terms: conditions — Nails, Ingrown

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evaluation of Apaisant Serum - Ingrown nails for Ingrown Toenails (Experimental): Subjects in this arm applied APAISANT SERUM - INGROWN NAILS topically to the affected nail area twice daily for 7 days. The serum provides a dual mechanical action: (1) lubrication of the nail plate with a lipid film to reduce friction with periungual tissue and (2) hydration of the nail to improve flexibility and prevent further irritation. The study was conducted as an open-label, before-and-after investigation, assessing changes in pain, discomfort, and clinical symptoms associated with ingrown toenails.
  Interventions: Device: APAISANT SERUM - INGROWN NAILS

INTERVENTIONS:
Device: APAISANT SERUM - INGROWN NAILS — Topical application of APAISANT SERUM - INGROWN NAILS twice daily for 7 days.

SUMMARY:
To open-label clinical study aims to evaluate the efficacy and safety of APAISANT SERUM - INGROWN NAILS, a Class IIa CE-marked medical device, in relieving pain and discomfort associated with inflamed ingrown nails. The study includes 22 subjects with ingrown nails at stage 1 or 2, who will apply the product twice daily for 7 days. The primary objective is to assess the reduction of pain using a Numerical Rating Scale (NRS, 0-10). Secondary objectives include assessing discomfort, inflammation, and overall symptom improvement. The study also evaluates investigator and patient global assessments, tolerance, and acceptability of the product. Safety will be monitored through clinical assessments and the collection of adverse events.

DETAILED DESCRIPTION:
This open-label, before-and-after study aims to assess the efficacy and tolerance of APAISANT SERUM - INGROWN NAILS in relieving pain, discomfort, and inflammation associated with ingrown toenails (stage 1 and 2). The study will include 22 subjects, ensuring a minimum of 20 analyzable cases. Participants will apply the product twice daily for 7 days at home.

Primary Objective:

To evaluate the reduction in pain at Day 7 (Visit 2) compared to baseline (Day 0), using a 0-10 Numerical Rating Scale (NRS).

Secondary Objectives:

To assess the reduction of discomfort at Day 7. To evaluate improvement in clinical symptoms (redness, edema, inflammation) and subjective symptoms (pain while touching, irritation).

To track daily pain and discomfort reduction from Day 1 to Day 7 compared to baseline.

To conduct Investigator Global Assessment (IGA) and Patient Global Assessment (PGA) at Day 7.

To assess subjective product acceptability, efficacy, and tolerance using a questionnaire.

To evaluate safety through clinical assessments, investigator evaluations, and monitoring of adverse events.

Study Design:

Participants will be enrolled based on inclusion and exclusion criteria, ensuring that subjects with stage 3 or 4 ingrown nails (with wounds, bleeding, or granulation tissue) are excluded. Data will be collected via investigator assessments and subject-reported outcomes.

Endpoints:

Primary Endpoint: Change in pain score after 7 days of treatment. Secondary Endpoints: Changes in discomfort, symptom improvement, pain/discomfort trajectory from Day 1 to Day 7, IGA, PGA, product tolerance, and safety (including adverse events).

Product Information:

Reference/Name: APAISANT SERUM - INGROWN NAILS Class: Class IIa CE-marked medical device Form: Liquid Dosage: Twice daily Duration: 7 days Administration Route: Topical application

Randomization and Blinding:

Not applicable; the study is open-label, with neither the investigator nor the subjects blinded to treatment.

Study Duration per Subject:

7 days The study aims to provide clinical evidence supporting the efficacy and tolerance of APAISANT SERUM - INGROWN NAILS in alleviating pain and discomfort from ingrown nails.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient having given her/his informed, written consent. 2. Patient cooperative and aware of the modalities of use and the necessity and duration of the controls so that perfect adhesion to the protocol can be expected.

  3. Patient being psychologically able to understand information and to give their/his/her consent.

  4. Male or female more than 3 years old. 5. Minor whose legally designated representative have given their free and express informed consent.

  6. Subject affiliated to a health social security system. 7. Female of childbearing potential should use a contraceptive regimen recognized as effective since at least 12 weeks before screening visit, during all the study and at least 1 month after the study end.

  8. Subjects presenting an inflamed Ingrown nails (folds) and with pain ;.
* state 1 : inlaid nail OR
* state 2 : peri inguale inflammation

Exclusion Criteria:

* 1. Subject presenting state 3 or 4 of the ingrown nails (presenting wounds, bleeding, discharge, granulation tissue growth).

  2. Subject who is currently participating, in another clinical study liable to interfere with the study assessments according to the investigator's assessment 3. Subject unable to understand the information given including study procedures (for linguistic or psychiatric reasons) and to give his/her consent in writing or to report required information in writing in his/her diary 4. Subject who, in the judgement of the investigator, is not likely to be compliant with study-related constraints and requirements 5. Subject who has forfeited his/her freedom by administrative or legal award or is under guardianship 6. For woman of childbearing potential: pregnant or breastfeeding or planning to get pregnant during the study 7. Subject having a skin disease, skin abnormalities, or dermatological condition on the studied area liable to interfere with the study assessments 8. Subject with a known history of allergy or contact dermatitis caused by any of the ingredients of the tested product 9. Acute, chronic or progressive disease or medical history considered by the investigator hazardous for the subject or incompatible with the study or liable to interfere with the study assessments 10. Any systemic treatment incompatible with the study or liable to interfere with the study assessments according to the investigator, in the weeks prior to the inclusion visit, ongoing or planned to be started during the study 11. Any topical treatment on the tested area incompatible with the study or liable to interfere with the study assessments according to the investigator, in the weeks prior to the inclusion visit, ongoing or planned to be started during the study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Change in pain severity of the ingrown toenail | Day 7 (D7) compared to baseline (D0)
  Pain severity will be assessed using the Numerical Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicate a worse outcome. The primary objective is to determine the effectiveness of Apaisant Serum - Ingrown Nails in reducing pain after 7 days of treatment.

SECONDARY OUTCOMES:
Change in discomfort severity of the ingrown toenail | Day 7 (D7) compared to baseline (D0)
  Discomfort severity will be measured using the Numerical Rating Scale (NRS), ranging from 0 (no discomfort) to 10 (worst possible discomfort). Higher scores indicate a worse outcome.
Improvement in ingrown nail symptom - redness | Day 7 (D7) compared to baseline (D0)
  Redness will be assessed using a 0-10 point Numerical Rating Scale (NRS), where 0 indicates no redness and 10 indicates the most severe redness. Higher scores indicate a worse outcome.
Improvement in ingrown nail symptom - edema | Day 7 (D7) compared to baseline (D0)
  Edemawill be assessed using a 0-10 point Numerical Rating Scale (NRS), where 0 indicates no edema and 10 indicates the most severe edema. Higher scores indicate a worse outcome.
Improvement in ingrown nail symptoms - inflammation | Day 7 (D7) compared to baseline (D0)
  Inflammation will be assessed using a 0-10 point Numerical Rating Scale (NRS), where 0 indicates no inflammation and 10 indicates the most severe inflammation. Higher scores indicate a worse outcome.
Improvement in ingrown nail symptoms - pain touch | Day 7 (D7) compared to baseline (D0)
  Pain on touch will be assessed using a 0-10 point Numerical Rating Scale (NRS), where 0 indicates no pain on touch and 10 indicates the most severe pain on touch. Higher scores indicate a worse outcome.
Improvement in ingrown nail symptoms - irritation | Day 7 (D7) compared to baseline (D0)
  Irritation will be assessed using a 0-10 point Numerical Rating Scale (NRS), where 0 indicates no irritation and 10 indicates the most severe irritation. Higher scores indicate a worse outcome.
Improvement in ingrown nail symptoms - overall appearance of the nails | Day 7 (D7) compared to baseline (D0)
  The overall appearance of the nails will be assessed using a 0-10 Numerical Rating Scale (NRS), where 0 indicates an unhealthy-looking nail and 10 indicates a completely healthy-looking nail. Higher scores indicate a better outcome.
Improvement in ingrown nail symptoms - gloss appearance of the nail | Day 7 (D7) compared to baseline (D0)
  Gloss appearance of the nail will be assessed using a 0-10 Numerical Rating Scale (NRS), where 0 indicates a dull nail and 10 indicates a very glossy nail. Higher scores indicate a better outcome.
Improvement in ingrown nail symptoms - nail smoothness | Day 7 (D7) compared to baseline (D0)
  Nail smoothness will be assessed using a 0-10 Numerical Rating Scale (NRS), where 0 indicates a rough nail and 10 indicates a very smooth nail. Higher scores indicate a better outcome.
Improvement in ingrown nail symptoms - the softness of the nail and its contour | Day 7 (D7) compared to baseline (D0)
  The softness of the nail and its contour will be assessed using a 0-10 Numerical Rating Scale (NRS), where 0 indicates a tough, callous nail and contour, and 10 indicates a soft nail and contour. Higher scores indicate a better outcome.
Improvement in ingrown nail symptoms - nail nourishment | Day 7 (D7) compared to baseline (D0)
  Nail nourishment will be assessed using a 0-10 Numerical Rating Scale (NRS), where 0 indicates a dry, weak, unnourished nail and 10 indicates a very nourished nail. Higher scores indicate a better outcome.
Change in pain over time | From Day 1 (D1) to Day 7 (D7) compared to baseline (D0)
  Pain levels will be recorded daily by participants using the Numerical Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicate a worse outcome.
Change in discomfort over time | From Day 1 (D1) to Day 7 (D7) compared to baseline (D0)
  Discomfort levels will be recorded daily by participants using the Numerical Rating Scale (NRS), ranging from 0 (no discomfort) to 10 (worst possible discomfort). Higher scores indicate a worse outcome.
Investigator Global Assessment (IGA) Score | Day 7 (D7)
  The investigator will evaluate overall improvement using a standardized clinical assessment scale ranging from -1 (worse) to 3 (very good improvement). Higher scores indicate a better outcome.
Patient Global Assessment (PGA) Score | Day 7 (D7)
  Participants will provide their own global assessment of improvement using a standardized scale ranging from -1 (worse) to 3 (very good improvement). Higher scores indicate a better outcome.
Subjective evaluation of general appreciation of the product | Day 7 (D7)
  Participants will rate their general appreciation of the product and its properties on a scale from 1 (very unpleasant) to 5 (very pleasant).
Subjective evaluation of efficacy | Day 7 (D7)
  Participants will indicate their level of agreement with statements regarding product effectiveness on a scale from 1 (strongly disagree) to 5 (strongly agree).
Subjective evaluation of future use of the product | Day 7 (D7)
  Participants will answer Yes or No to questions about their intention to use the product in the future.
Tolerance and safety assessment | Throughout the study (D0-D7)
  Any adverse events (AEs) will be collected and analyzed to evaluate the safety profile of the investigational device throughout the study.
Illustrative macrophotographs | Day 0 (D0) and Day 7 (D7)
  Standardized images will be taken to document the visual improvement of the ingrown toenail condition throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Dermscan Poland, Gdansk, Poland, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing plans have not yet been finalized. A decision will be made later.